CLINICAL TRIAL: NCT01250912
Title: Three Dimension Neuron Imaging Using 123I-metaiodobenzylguanidine Single Photon Emission Computed Tomography to Guide Ventricular Tachycardia Ablations
Brief Title: Imaging With a Radio Tracer to Guide VT Ablations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Timm-Michael Dickfeld, Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00043324
Record Dates: First submitted 2010-07-28; First posted 2010-12-01 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Ventricular Tachycardia; Arrhythmia
Keywords: Ablation; Arrythmia; Imaging
MeSH Terms: conditions — Tachycardia, Ventricular; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imaging Tracer (Experimental): No arms, the Radio tracer will be used in all subjects imaging tests.
  Interventions: Drug: 123I-metaiodobenzylguanidine

INTERVENTIONS:
Drug: 123I-metaiodobenzylguanidine — FDA Approved for use in Cancer patients. This use is Off Label. For the imaging study, an activity of 370 MBq (10 mCi) 123I-mIBG (GE Healthcare) will be administered intravenously, and a 10-minute planar image of the anterior thorax (128_128 matrix) will be acquired beginning 15 minutes after tracer injection.
  Other Names: MIGB

SUMMARY:
Some patients are at risk for life-threatening fast heart rates. These can frequently be treated by using a catheter inside the heart to burn away the cells that create the fast heart rates. The purpose of this study is to image the nerves inside the heart of those patients. The investigators want to find out if abnormalities in the nervous system in the heart can help the physician to find the area that needs to be burnt away.

DETAILED DESCRIPTION:
Ventricular tachycardia is the next frontier in cardiology. Patients that have scar in the heart (for example after heart attacks) are at an increased risk of developing ventricular tachycardia. In these patients ventricular tachycardia represents an electrical wave front that circulates in the heart muscle using the scar in the heart. An increasing number of patients with ventricular tachycardia require cauterization (burning away) of the tissue to treat this life-threatening condition. The goal of this cauterization or ablation is to destroy "highways of surviving tissue" inside the scar, that allow ventricular tachycardia to exist. However, this can be very lengthy procedure (>5 hours) that has only a moderate success in the long run. Therefore, new treatment approaches are needed to make this procedure better.

The purpose of this study is to assess if radio tracers showing the nerve distribution in the heart (cardiac innervation) can be used in addition to the current technology ("voltage mapping") to identify the area that needs to be ablated (burnt away) to treat life-threatening fast heart rates (ventricular tachycardia)

Certain patterns of nerve distribution in the heart (sympathetic cardiac innervation) have been shown to predict outcome for different heart diseases, like heart transplant, coronary artery disease, heart failure, arrhythmias. One substance that allows visualization of the cardiac innervation is 123I-metaiodobenzylguanidine (123I-MIBG), which could provide additional information to understand and treat ventricular tachycardia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ventricular arrhythmias requiring VT Ablation
* Patients must be 18 years of age or older
* Patient must be able to sign consent form
* Patient must be willing to come back for the 6 month visit for additional study procedures

Exclusion Criteria:

* Patient under 18 years old
* Inability to sign consent
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timm R Dickfeld, MD,Ph.D, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, EP Lab, Rm. N3W77, Baltimore, Maryland, United States

REFERENCES:
- [Background] Tian J, Smith MF, Jeudy J, Dickfeld T. Multimodality fusion imaging using delayed-enhanced cardiac magnetic resonance imaging, computed tomography, positron emission tomography, and real-time intracardiac echocardiography to guide ventricular tachycardia ablation in implantable cardioverter-defibrillator patients. Heart Rhythm. 2009 Jun;6(6):825-8. doi: 10.1016/j.hrthm.2009.02.032. Epub 2009 Feb 24. No abstract available. PMID 19467512
- [Background] Tian J, Smith MF, Chinnadurai P, Dilsizian V, Turgeman A, Abbo A, Gajera K, Xu C, Plotnick D, Peters R, Saba M, Shorofsky S, Dickfeld T. Clinical application of PET/CT fusion imaging for three-dimensional myocardial scar and left ventricular anatomy during ventricular tachycardia ablation. J Cardiovasc Electrophysiol. 2009 Jun;20(6):567-604. doi: 10.1111/j.1540-8167.2008.01377.x. PMID 19207761
- [Background] Dickfeld T, Kocher C. The role of integrated PET-CT scar maps for guiding ventricular tachycardia ablations. Curr Cardiol Rep. 2008 Mar;10(2):149-57. doi: 10.1007/s11886-008-0025-1. PMID 18417016
- [Result] Klein T, Abdulghani M, Smith M, Huang R, Asoglu R, Remo BF, Turgeman A, Mesubi O, Sidhu S, Synowski S, Saliaris A, See V, Shorofsky S, Chen W, Dilsizian V, Dickfeld T. Three-dimensional 123I-meta-iodobenzylguanidine cardiac innervation maps to assess substrate and successful ablation sites for ventricular tachycardia: feasibility study for a novel paradigm of innervation imaging. Circ Arrhythm Electrophysiol. 2015 Jun;8(3):583-91. doi: 10.1161/CIRCEP.114.002105. Epub 2015 Feb 23. PMID 25713216

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Receiving MIBG Imaging: All patients received MIBG imaging before and 6 months after VT ablation
Period: Overall Study
Arm/Group | Patients Receiving MIBG Imaging
Started | 20
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- MIBG Imaging on Top of Standard of Care VT Ablation: MIBG/SPECT imaging prior to, and 6 months after the ablation. 123I-metaiodobenzylguanidine: FDA Approved for use in Cancer patients. This use is Off Label. For the imaging study, an activity of 370 MBq (10 mCi) 123I-mIBG (GE Healthcare) will be administered intravenously, and a 10-minute planar image of the anterior thorax (128_128 matrix) will be acquired beginning 15 minutes after tracer injection.
Arm/Group | MIBG Imaging on Top of Standard of Care VT Ablation
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Ejection Fraction [Mean (Standard Deviation); unit: percent of LV ejection fraction] | 12.3 (25.2)
Comorbidities [Count of Participants; unit: Participants]
  Diabetes Mellitus | 6
  Hypertension | 16
  Hyperlipidemia | 12
  Atrial Fibrillation | 7
NYHA Heart Class [Count of Participants; unit: Participants]
  NYHA I (Asymptomatic) Best category | 0
  NYHA II (Dyspnea on severe activity) | 7
  NYHA III (Dyspnea on ordinary activity | 11
  NYHA IV (Dyspnea at rest) Worst category | 2

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Percentage of Patients With Scar in Each Segment as Determined by MIBG SPECT Versus Electroanatomic at Baseline
Description: Scar Measurement on both MIBG 3D map and electroanatomic scare defined as bipolar voltage <0.5mV using Standard 17-segment American Heart Association areas.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- MIBG/SPECT: Assessment by MIBG/SPECT
- Electroanatomic Imaging Assessment: Assessment electroanatomic by a bipolar voltage of <0.5 mV.
Arm/Group | MIBG/SPECT | Electroanatomic Imaging Assessment
Number analyzed (Participants) | 20 | 20
Participants
  Basal Anterior | 2 | 4
  basal Anteroseptal | 1 | 4
  Basal Inferoseptal | 11 | 9
  Basal Inferior | 18 | 10
  Basal Anterolateral | 16 | 13
  Mid Anterior | 2 | 6
  Mid Anteroseptal | 3 | 6
  Mid Inferoseptal | 14 | 11
  Mid Inferior | 15 | 13
  Mid Inferolateral | 13 | 10
  Mid Anterolateral | 3 | 4
  Apical Anterior | 2 | 4
  Apical Septal | 12 | 9
  Apical Inferior | 14 | 11
  Apical Lateral | 11 | 8
  Apex | 11 | 8

2. Secondary Outcome: Median Segmental MIBG Uptake at Baseline
Description: The median uptake of the standard 17 heart segments was determined at baseline
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: percentage of maximum uptake
Groups:
- MIBG Imaging at Baseline: MIBG/SPECT imaging prior to the ablation. 123I-metaiodobenzylguanidine: For the imaging study, an activity of 370 MBq (10 mCi) 123I-mIBG (GE Healthcare) was administered intravenously, and a 10-minute planar image of the anterior thorax (128_128 matrix) was acquired beginning 15 minutes after tracer injection.
Arm/Group | MIBG Imaging at Baseline
Number analyzed (Participants) | 19
percentage of maximum uptake | 52 [50 to 62]

3. Secondary Outcome: Median Segmental MIBG Uptake at 6 Months After Ablation
Description: MIBG/SPECT imaging 6 months after ablation. 123I-metaiodobenzylguanidine: For the imaging study, an activity of 370 MBq (10 mCi) 123I-mIBG (GE Healthcare) was administered intravenously, and a 10-minute planar image of the anterior thorax (128_128 matrix) was acquired beginning 15 minutes after tracer injection.
Time Frame: 6 months after ablation
Measure: Mean (Inter-Quartile Range); unit: percentage of maximum uptake
Groups:
- MIBG Imaging at 6 Months: MIBG/SPECT imaging 6 months after ablation. 123I-metaiodobenzylguanidine: For the imaging study, an activity of 370 MBq (10 mCi) 123I-mIBG (GE Healthcare) was administered intravenously, and a 10-minute planar image of the anterior thorax (128_128 matrix) was acquired beginning 15 minutes after tracer injection.
Arm/Group | MIBG Imaging at 6 Months
Number analyzed (Participants) | 19
percentage of maximum uptake | 48 [46 to 56]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Clinicaltrials.gov definitions were used
Groups:
- MIBG Imaging on Top of Standard of Care VT Ablation: MIBG/SPECT imaging prior to, and 6 months after the ablation. For the imaging study, an activity of 370 MBq (10 mCi) 123I-mIBG (GE Healthcare) will be administered intravenously, and a 10-minute planar image of the anterior thorax (128_128 matrix) will be acquired beginning 15 minutes after tracer injection.
Arm/Group | MIBG Imaging on Top of Standard of Care VT Ablation
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIBG Imaging on Top of Standard of Care VT Ablation (N=20)
Death due to unrelated non cardiac cause (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-09-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT01250912/Prot_SAP_000.pdf